CLINICAL TRIAL: NCT01434602
Title: A Phase I-II Trial of Everolimus and Sorafenib in Patients With Recurrent High-Grade Gliomas
Brief Title: Phase I-II Everolimus and Sorafenib in Recurrent High-Grade Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Gilbert, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160011; 16-C-0011
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Brain Tumor; Glioblastoma; Anaplastic Glioma
Keywords: Chemotherapy; Brain Tumor; Glioblastoma; Anaplastic Glioma
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma | interventions — Everolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase I (Experimental): Daily everolimus (days 1- 28) in combination with sorafenib as per the Phase I dosing table. Maximum tolerated dose. Dose Escalation.
  Interventions: Drug: everolimus; Drug: sorafenib
- 2/Phase II (Experimental): Combination of sorafenib and everolimus. Sorafenib 400mg twice daily will be taken for 7 days on, then 7 days off. Everolimus 5mg will be taken daily. Determined from dose escalation in phase I, maximum tolerated dose -1.
  Interventions: Drug: everolimus; Drug: sorafenib

INTERVENTIONS:
Drug: everolimus — Patients will be treated with daily everolimus (days 1-28) in combination with sorafenib; There is not a defined set maximum number of cycles that a patient may have; Phase I Dose Escalation: 5mg to 10mg daily.
  Other Names: Zortress
Drug: sorafenib — Patients will be treated with sorafenib in combination with everolimus (days 1-28); There is not a defined set maximum number of cycles that a patient may have; Phase I Dose Escalation 400mg-600mg twice a day (bid) or 400mg-800mg twice a day, 7 days on and 7 days off.
  Other Names: Nexavar

SUMMARY:
The goal of Phase 1 of this clinical research study is to find the highest tolerable dose and best schedule of the combination of everolimus and sorafenib that can be given to patients with malignant glioma.

The goal of Phase 2 of this study to learn if the combination of everolimus and sorafenib can help to control malignant glioma. The safety of this combination will also be studied in both phases.

DETAILED DESCRIPTION:
Background

* Although malignant gliomas display genetic heterogeneity, several key proliferation and survival signaling pathways have been identified.
* Recent work has focused on targeting these tumor specific pathways in hopes of improving treatment efficacy and minimizing treatment toxicity. Because molecularly targeted agents have been mostly ineffective when used alone, combination therapy that inhibits multiple pathways is an appealing strategy.
* Sorafenib is an oral multi-kinase inhibitor with effects on tumor proliferation and tumor angiogenesis. Although most GBMs lack rapidly accelerated fibrosarcoma (RAF) mutations, targeting the RAF/methyl ethyl ketone (MEK)/extracellular-signal-regulated kinase (ERK) pathway may be beneficial as this pathway may be activated by other genetic alterations upstream from RAF.
* The mammalian target of rapamycin (mTOR) protein is a downstream component of the Phosphoinositide 3-kinases (PI3K)/Protein kinase B (Akt) pathway. Everolimus (everolimus; Novartis) is a novel oral derivative of rapamycin.
* Combining everolimus and sorafenib allows targeting of both the PI3K pathway and the RAF-MAPK pathway and in addition targets vascular endothelial growth factor (VEGF) and platelet-derived growth factor (PDGF), other active targets in malignant glioma.

Objectives

Phase 1

-To determine the maximum tolerated dose and safety of everolimus in combination with

sorafenib for patients with recurrent malignant gliomas.

Phase 2

* 6 months progression free survival rate for glioblastoma patients with no prior bevacizumab exposure treated with everolimus and sorafenib at the maximum tolerated dose as determined in the phase I study.
* 3 months progression free survival rate for glioblastoma patients with prior bevacizumab exposure treated with everolimus and sorafenib at the maximum tolerated dose as determined in the phase I study.
* 6 months progression free survival rate for Anaplastic Glioma (AG) patients with no prior bevacizumab exposure treated with everolimus and sorafenib at the maximum tolerated dose as determined in the phase I study.

Eligibility

* Patients with histologically proven recurrent intracranial malignant glioma will be eligible for the phase I/II component of this protocol.
* Patients must be >= 18 years old with a Karnofsky performance status of greater than or equal to 60
* No more than 2 prior chemotherapies and 1 relapse. Prior bevacizumab therapy is allowed.

Design

* This is a phase 1 /2 study of everolimus and sorafenib in patients with recurrent high-grade gliomas.
* Phase 1: Patients will be treated with daily everolimus (days 1-28) in combination with sorafenib.
* Phase 2: Patients will be treated with the combination of sorafenib and everolimus. Sorafenib will be taken daily for 7 days on, then 7 days off. Everolimus will be taken daily.
* There is not a defined set maximum number of cycles that a patient may have. Patients may continue with protocol therapy until criteria for Off Treatment is met. Patients will then be followed every 3 months for survival status.
* There will be an accrual of approximately 3-6 eligible patients per cohort to the Phase I component of the study. Patients removed at any time for toxicity are evaluable. Phase I patients removed from study treatment within 28 days for reasons other than toxicity may be replaced.
* There will be a total accrual of approximately 82 eligible patients to the Phase II study (34 recurrent GBM with no prior exposure to bevacizumab, 16 recurrent Anaplastic Glioma with no prior exposure to bevacizumab, and 32 glioblastoma with prior exposure to bevacizumab).

ELIGIBILITY:
* INCLUSION CRITERIA:

General Inclusion Criteria

1. Patients with histologically proven recurrent intracranial malignant glioma will be eligible for the phase I/II component of this protocol. Malignant glioma includes glioblastoma (GBM), Gliosarcoma (GS), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma not otherwise specified (NOS) (not otherwise specified). Patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a malignant glioma is made.
2. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must have signed an authorization for the release of their protected health information at all sites except the National Institutes of Health (NIH).
3. Patients must be greater than or equal to 18 years old.
4. Patients must have a Karnofsky performance status of greater than or equal to 60.
5. No more than 2 prior chemotherapies and 1 relapse. Prior bevacizumab therapy is allowed.

   -Patients must have recovered from the toxic effects of prior therapy: >3 weeks for biologic therapies or non-cytotoxic therapies, >4 weeks for cytotoxic therapies, and >6 weeks for nitrosoureas. Any questions related to the definition of non- cytotoxic agents should be directed to the Study Chair.

   NOTE: 13 cis-retinoic acid (Accutane) as biologic therapy has a washout period of 14 days.
6. Patients must have adequate bone marrow function (white blood cell (WBC) >= 3.0 x 10^9/L, absolute neutrophil count (ANC) >= 1.5 X 10^9/L, platelet count of >=100 x 10^9/L, and hemoglobin >= 10 gm/dL), adequate liver function (Serum glutamic oxaloacetic transaminase (SGOT) and bilirubin < 2 times upper limit of normal (ULN), and adequate renal function (creatinine < 1.7mg/dL or creatinine clearance greater than or equal to 60 cc/min) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.
7. Patients must have shown unequivocal radiographic evidence for tumor progression by magnetic resonance imaging (MRI) or computed tomography (CT) scan. A scan should be performed within 14 days prior to registration and on a steroid dose that has been stable or decreasing for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MRI/CT is required. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement. Measurable disease is NOT required.

   Note: MRI is the preferable imaging method; CT scan may be used in cases where an MRI cannot be obtained.
8. Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

   * They have recovered from the effects of surgery and be > 3 weeks from surgery.
   * Residual disease following resection of recurrent malignant glioma is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/ MRI should be done no later than 96 hours in the immediate post-operative period or at least 4 weeks post-operatively, within 14 days prior to registration. If the 96-hour scan is more than 14 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.
9. Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 12 weeks from the completion of radiation therapy to registration; except if patients underwent surgery within 12 weeks and pathology is consistent with recurrent tumor.
10. Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon either positron emission tomography (PET) or Thallium scanning, magnetic resonance (MR) spectroscopy or surgical/pathological documentation of disease.
11. Women of childbearing potential must have a negative beta human chorionic gonadotropin (B-HCG) pregnancy test documented within 7 days prior to taking the first dose of study medications.
12. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the international normalized ratio (INR) should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.

Phase I Inclusion Criteria:

The following modifications to the general eligibility criteria apply to Phase I patients only.

-Patients may have had treatment for any number of prior relapses. Relapse is defined as progression following initial therapy (i.e., surgery and radiation+/- chemo if that was used as initial therapy).

Phase II Inclusion Criteria:

Phase II patients must meet the following Eligibility Criteria in addition to the General Criteria described above.

* Patients may have had treatment for no more than 1 prior relapse (i.e., failed 2 lines of treatment-initial therapy and therapy for first relapse) at 2nd relapse, treatment per BTTC09-01 is an option. Relapse is defined as progression following initial therapy (i.e., radiation+/- chemo if that was used as initial therapy). The intent therefore is that patients had no more than 2 prior therapies (initial and treatment for 1 relapse). If the patient had a surgical resection for relapsed disease and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered as 1 relapse. For patients who had prior therapy for a low-grade glioma, the surgical diagnosis of a high-grade glioma will be considered the first relapse.
* Patients must not have received prior therapy with sorafenib, everolimus, or related drugs such as tyrosine kinase inhibitors, vascular endothelial growth factor (VEGF) inhibitors (except bevacizumab), or mTOR inhibitors.

EXCLUSION CRITERIA:

General Exclusion Criteria

1. Patients has any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
2. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
3. Patients has an active infection or serious intercurrent medical illness.
4. Patients has any disease that will obscure toxicity or dangerously alter drug metabolism.
5. Patients must not be on enzyme inducing anti-convulsants. If patients were previously on enzyme-inducing antiepileptic drugs (EIAEDs) and these have been discontinued, patients must have been off the agent for at least 2 weeks prior to first study drug administration. For patients who need to start an AED, or the AED needs to be changed, it is strongly recommended that all efforts should be made to use a non-EIAED.
6. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: Symptomatic congestive heart failure of New York heart Association Class III or IV unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug or any other clinically significant cardiac disease severely impaired lung function as defined as spirometry and diffusing capacity for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN, active (acute or chronic) or uncontrolled severe infections, liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
7. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
8. Uncontrolled hypertension defined as systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
9. Known human immunodeficiency virus (HIV) infection or chronic or acute Hepatitis B or C. Note: Patients who have a history of hepatitis B virus (HBV) and HCB infection are eligible, however, they must receive prophylactic antiviral therapy for 1-2 weeks prior to receiving study drug
10. Thrombolic or embolic events (except deep vein thrombosis (DVT) or pulmonary embolus) such as a Cerebrovascular accident including transient ischemic attacks within the past 6 months.
11. Pulmonary hemorrhage/bleeding event greater than or equal to Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 within 4 weeks of first dose of study drug.
12. Any other hemorrhage/bleeding event greater than or equal to CTCAE Grade 3 within 4 weeks of first dose of study drug.
13. Serious non-healing wound, non-healing ulcer, or bone fracture.
14. Evidence or history of bleeding diathesis or coagulopathy
15. Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
16. Use of St. John's Wort, or rifampin (rifampicin), or other strong Cytochrome P450 3A4 (CYP34A) inducers. Dexamethasone is okay as long as the dose is 16 mg /day or less.

    Note: Patients who are on the above referenced medications may be considered eligible with a washout period of 14 days. Contact the coordinating center to discuss patients with the above aforementioned agents before patient registration.
17. Known or suspected allergy to sorafenib, everolimus, or any agent given in the course of this trial.
18. Any condition that impairs patient's ability to swallow whole pills.
19. Any malabsorption problem.
20. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
21. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Barrier contraceptives must be used throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of everolimus and sorafenib).
22. Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
23. Patients with a known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus) or to its excipients.
24. History of noncompliance to medical regimens.
25. Patients unwilling to or unable to comply with the protocol.
26. Patients on total daily dose of dexamethasone greater than 16 mg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-10-02 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2021-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Gilbert, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0011.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study started at MD Anderson under Dr. Gilbert in 2012 and transferred to the National Cancer Institute (NCI).
Groups:
- Phase I Dose Level I Sorafenib 400mg Twice Daily + Everolimus 5mg Daily: Phase I Dose Level 1 Dose Escalation Participants with recurrent malignant glioma, with or without prior exposure to bevacizumab will be treated with Sorafenib 400mg twice daily + Everolimus 5 mg daily by mouth (days 1-28). There is not a defined set maximum number of cycles that a patient may have.
- Phase I Dose Level -1 Sorafenib 400mg Twice Daily, 7 Days on, 7 Off + Everolimus 5mg Daily: Phase I Dose Level -1 Dose Escalation Phase Participants with recurrent malignant glioma, with or without prior exposure to bevacizumab will be treated with Sorafenib 400mg twice daily 7 days on, 7 days off + Everolimus 5 mg daily by mouth (days 1-28). There is not a defined set maximum number of cycles that a patient may have. Sorafenib will be given on days 1-7 and days 15-21.
- Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily: Phase 2 Recommended Phase 2 Dose Recurrent glioblastoma with no prior exposure to bevacizumab Participants will be treated with Sorafenib 400mg twice daily 7 days on, 7 days off + Everolimus 5 mg daily by mouth (days 1-28). There is not a defined set maximum number of cycles that a patient may have. Sorafenib will be given on days 1-7 and days 15-21.
- Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily: Phase 2 Recommended Phase 2 Dose Recurrent glioblastoma with prior exposure to bevacizumab Participants will be treated with Sorafenib 400mg twice daily 7 days on, 7 days off + Everolimus 5 mg daily by mouth (days 1-28). There is not a defined set maximum number of cycles that a patient may have.
  Sorafenib will be given on days 1-7 and days 15-21.
- Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily: Phase 2 recommended phase 2 dose Participants with Anaplastic Glioma with no prior exposure to bevacizumab (Grade III Glioma Group) will be treated with Sorafenib 400mg twice daily 7 days on, 7 days off + Everolimus 5 mg daily by mouth (days 1-28). There is not a defined set maximum number of cycles that a patient may have. Sorafenib will be given on days 1-7 and days 15-21.
Period: Phase I Dose Escalation
Arm/Group | Phase I Dose Level I Sorafenib 400mg Twice Daily + Everolimus 5mg Daily | Phase I Dose Level -1 Sorafenib 400mg Twice Daily, 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
Started | 6 | 7 | 0 | 0 | 0
Completed | 6 | 6 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Participant was underdosed (i.e., was taking incorrect dose at home)/Not evaluable | 0 | 1 | 0 | 0 | 0
Period: Phase II Recommended Phase 2 Dose
Arm/Group | Phase I Dose Level I Sorafenib 400mg Twice Daily + Everolimus 5mg Daily | Phase I Dose Level -1 Sorafenib 400mg Twice Daily, 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
Started | 0 | 0 | 12 | 40 | 21
Completed | 0 | 0 | 12 | 31 | 19
Not Completed | 0 | 0 | 0 | 9 | 2
Not completed — Active progression before start of treatment | 0 | 0 | 0 | 1 | 0
Not completed — Bilateral large pulmonary embolisms in the right and left main pulmonary arteries | 0 | 0 | 0 | 1 | 0
Not completed — Started new therapy | 0 | 0 | 0 | 1 | 0
Not completed — Decline in patient condition/health/ADL's | 0 | 0 | 0 | 1 | 0
Not completed — Transfer of care | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1
Not completed — Switched to alternative treatment | 0 | 0 | 0 | 1 | 0
Not completed — Refused further treatment | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on 7 Off + Everolimus 5mg Daily: Phase 2 Recommended Phase 2 Dose Recurrent glioblastoma with no prior exposure to bevacizumab Participants will be treated with Sorafenib 400mg twice daily 7 days on, 7 days off + Everolimus 5 mg daily by mouth (days 1-28). There is not a defined set maximum number of cycles that a patient may have. Sorafenib will be given on days 1-7 and days 15-21.
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level I Sorafenib 400mg Twice Daily + Everolimus 5mg Daily | Phase I Dose Level -1 Sorafenib 400mg Twice Daily, 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on 7 Off + Everolimus 5mg Daily | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Total
Number analyzed (Participants) | 6 | 7 | 12 | 40 | 21 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 10 | 34 | 19 | 74
  >=65 years | 0 | 2 | 2 | 6 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.90 (12.80) | 48.65 (19.32) | 51.34 (12.13) | 51.74 (14.34) | 44.09 (14.43) | 49.23 (14.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 5 | 16 | 8 | 31
  Male | 5 | 6 | 7 | 24 | 13 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 1 | 2 | 0 | 3
  White | 5 | 6 | 10 | 37 | 18 | 76
  Unknown | 1 | 1 | 0 | 1 | 3 | 6
  Other | 0 | 0 | 1 | 0 | 0 | 1
  Missing Ethnicity | 6 | 7 | 12 | 27 | 19 | 71
  Hispanic | 0 | 0 | 0 | 0 | 2 | 2
  Not Hispanic | 0 | 0 | 0 | 13 | 0 | 13
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 12 | 40 | 21 | 86

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Everolimus for Participants With Recurrent Malignant Gliomas
Description: Maximum tolerated dose of everolimus for participants with recurrent malignant gliomas. MTD is defined as the dose at which fewer than one-third of participants experience a dose limiting toxicity (DLT) to one of the study drugs. A DLT is any grade 3 thrombocytopenia, grade 4 anemia, grade 4 neutropenia, or febrile neutropenia of any grade. Any non-hematologic grade 3 or grade 4 toxicity, excluding alopecia and/or hand/foot reaction. Failure to recover from toxicities (to grade 1 or less) to be eligible for re-treatment with everolimus within 14 days of the last dose of everolimus.
Time Frame: First 28 days of treatment only (cycle 1)
Measure: Number; unit: mg
Groups:
- All Participants: All participants with recurrent malignant glioma, with or without prior exposure to bevacizumab on phase I dose level 1 and phase I dose level-1.
  Phase I Dose Level 1: Sorafenib 400mg twice daily + Everolimus 5 mg daily by mouth (days 1-28).
  Phase I Dose Level -1:
  Sorafenib 400mg twice daily 7 days on, 7 days off + Everolimus 5 mg daily by mouth (days 1-28). Sorafenib will be given on days 1-7 and days 15-21.
  There is not a defined set maximum number of cycles that a participant may have.
Arm/Group | All Participants
Number analyzed (Participants) | 13
mg | 5

2. Primary Outcome: Maximum Tolerated Dose of Sorafenib for Participants With Recurrent Malignant Gliomas
Description: Maximum tolerated dose of sorafenib for participants with recurrent malignant gliomas. MTD is defined as the dose at which fewer than one-third of participants experience a dose limiting toxicity (DLT) to one of the study drugs. A DLT is any grade 3 thrombocytopenia, grade 4 anemia, grade 4 neutropenia, or febrile neutropenia of any grade. Any non-hematologic grade 3 or grade 4 toxicity, excluding alopecia and/or hand/foot reaction. Failure to recover from toxicities (to grade 1 or less) to be eligible for re-treatment with sorafenib within 14 days of the last dose of sorafenib.
Time Frame: First 28 days of treatment only (cycle 1)
Population: The dosing schedule for the MTD is 400mg twice a day (BID) 7 days on/7 days off.
Measure: Number; unit: mg
Arm/Group | All Participants
Number analyzed (Participants) | 13
mg | 400

3. Primary Outcome: Percentage of Participants Who Survived Without Disease Progression at 6 Months After Treatment for Glioblastoma Participants With no Prior Bevacizumab Exposure
Description: Percentage of participants who survived without disease progression at 6 months after treatment for glioblastoma participants with no prior bevacizumab exposure. Progression was measured by brain magnetic resonance imaging (MRI) tumor measurements. Progression is defined as >25% increase in the sum of products of perpendicular diameters of enhancing lesions (over baseline if no decrease) on stable or increasing dose of corticosteroids; and/or significant increase in T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR) non-enhancing lesion on stable or increasing doses of corticosteroids compared to baseline scan or best response following initiation or therapy, not due to co-morbid events (radiation therapy, demyelination, ischemic injury, infection, seizures, postoperative changes, or other treatment effects). Any new lesion.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
Number analyzed (Participants) | 12
Percentage of participants | 8.33 [0.51 to 31.1]

4. Primary Outcome: Percentage of Participants Who Survived Without Disease Progression at 3 Months After Treatment for Glioblastoma Participants With Prior Bevacizumab Exposure
Description: Percentage of participants who survived without disease progression at 3 months after treatment for glioblastoma participants with prior bevacizumab exposure. Progression was measured by brain magnetic resonance imaging (MRI) tumor measurements. Progression is defined as >25% increase in the sum of products of perpendicular diameters of enhancing lesions (over baseline if no decrease) on stable or increasing dose of corticosteroids; and/or significant increase in T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR) non-enhancing lesion on stable or increasing doses of corticosteroids compared to baseline scan or best response following initiation or therapy, not due to co-morbid events (radiation therapy, demyelination, ischemic injury, infection, seizures, postoperative changes, or other treatment effects). Any new lesion.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
Number analyzed (Participants) | 40
Percentage of participants | 12.9 [4.07 to 27.0]

5. Primary Outcome: Percentage of Participants Who Survived Without Disease Progression at 6 Months After Treatment for Anaplastic Glioma (AG) Participants With no Prior Bevacizumab Exposure
Description: Percentage of participants who survived without disease progression at 6 months after treatment for anaplastic glioma (AG) participants with no prior bevacizumab exposure. Progression was measured by brain magnetic resonance imaging (MRI) tumor measurements. Progression is defined as >25% increase in the sum of products of perpendicular diameters of enhancing lesions (over baseline if no decrease) on stable or increasing dose of corticosteroids; and/or significant increase in T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR) non-enhancing lesion on stable or increasing doses of corticosteroids compared to baseline scan or best response following initiation or therapy, not due to co-morbid events (radiation therapy, demyelination, ischemic injury, infection, seizures, postoperative changes, or other treatment effects). Any new lesion.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
Number analyzed (Participants) | 21
Percentage of participants | 26.7 [8.26 to 49.6]

6. Secondary Outcome: Median Amount of Time Participants Survives Without Disease Progression for Groups A, B, and C Treated With Everolimus and Sorafenib
Description: Median amount of time participants survives without disease progression for Groups A, B, and C treated with everolimus and sorafenib. Progression was measured by brain magnetic resonance imaging (MRI) tumor measurements. Progression is defined as >25% increase in the sum of products of perpendicular diameters of enhancing lesions (over baseline if no decrease) on stable or increasing dose of corticosteroids; and/or significant increase in T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR) non-enhancing lesion on stable or increasing doses of corticosteroids compared to baseline scan or best response following initiation or therapy, not due to co-morbid events (radiation therapy, demyelination, ischemic injury, infection, seizures, postoperative changes, or other treatment effects). Any new lesion.
Time Frame: Up to 6 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
Number analyzed (Participants) | 12 | 40 | 21
Months | 1.92 [.967 to 3.73] | 1.17 [.933 to 1.90] | 1.87 [.933 to 4.73]

7. Secondary Outcome: Objective Response for Participants With Recurrent Malignant Gliomas (Group A, Group B, and Group C) Treated With Everolimus and Sorafenib
Description: Objective response for participants with recurrent malignant gliomas treated with everolimus and sorafenib was assessed by brain magnetic resonance imaging (MRI) tumor measurements. Complete Response is complete disappearance of all CE measurable and evaluable disease. Partial Response is greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of the two largest CE measurable lesions, sustained for at least 4 weeks. Progressive Disease >25% increase in the sum of products of perpendicular diameters of enhancing lesions (over baseline if no decrease) on stable or increasing dose of corticosteroids, significant increase in T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR) non-enhancing lesion on stable or increasing doses of corticosteroids compared to baseline scan or best response following initiation or therapy, not due to co-morbid events, or any new lesion. Stable Disease does not qualify for CR, PR, or progression.
Time Frame: After 1 cycle of treatment, or those who exhibit objective progression prior the end of cycle 1 (one cycle = 28 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on 7 Off + Everolimus 5mg Daily | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
Number analyzed (Participants) | 12 | 40 | 21
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 2
  Progressive Disease | 4 | 17 | 7
  Stable Disease | 8 | 16 | 10
  Not Evaluable | 0 | 7 | 2

8. Secondary Outcome: Median Amount of Time a Participant Survives After Therapy for Participants With Recurrent Malignant Glioma (Group A, Group B, and Group C) Treated With Everolimus and Sorafenib Measured From the Time of Study Enrollment
Description: Median amount of time a participant survives after therapy for participants with recurrent malignant glioma (Group A, Group B, and Group C) treated with everolimus and sorafenib measured from the time of study enrollment.
Time Frame: From the time of study enrollment up to 1.5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
Number analyzed (Participants) | 12 | 40 | 21
Months | 7.75 [3.17 to 17.57] | 4.77 [2.77 to 6.53] | 11.97 [6.40 to 17.97]

9. Secondary Outcome: Rate of Participants Symptom Severity
Description: To evaluate the occurrence of symptoms and correlate to disease progression and tolerance to treatment using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) self-reporting tool. The MDASI-BT consists of 23 symptoms rated on an 11-point scale (0 - not present, to 10 - as bad as you can imagine) to indicate the presence and severity of the symptom. We calculated the mean core symptom severity at the time of clinical evaluation.
Time Frame: Completed at baseline, before a brain or spine magnetic resonance imaging (MRI)/clinical evaluation, and at cycle 1-2, cycle 4, cycle 6, cycle 8, cycle 10 and cycle 12 (each cycle is 28 days)
Population: 78/86 participants were evaluable for this outcome measure. 1 participant had active progression before start of treatment, 3 participants did not have data available (no confirmed treatment dates), and 4 participants were missing questionnaires, thus were not counted. 0 analyzed = Participants were taken off therapy before reaching the timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Phase 1 Dose LEvel 1 Sorafenib 400mg Twice Daily + Everolimus 5mg Daily: Phase I Dose Level 1 Dose Escalation Participants with recurrent malignant glioma, with or without prior exposure to bevacizumab will be treated with Sorafenib 400mg twice daily + Everolimus 5 mg daily by mouth (days 1-28). There is not a defined set maximum number of cycles that a patient may have.
- Phase 1 Dose Level -1 Sorafenib 400mg Twice Daily 7 Days On, & Days Off + Everolimus Daily: Phase I Dose Level -1 Dose Escalation Phase Participants with recurrent malignant glioma, with or without prior exposure to bevacizumab will be treated with Sorafenib 400mg twice daily 7 days on, 7 days off + Everolimus 5 mg daily by mouth (days 1-28). There is not a defined set maximum number of cycles that a patient may have. Sorafenib will be given on days 1-7 and days 15-21.
Arm/Group | Phase 1 Dose LEvel 1 Sorafenib 400mg Twice Daily + Everolimus 5mg Daily | Phase 1 Dose Level -1 Sorafenib 400mg Twice Daily 7 Days On, & Days Off + Everolimus Daily | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on 7 Off + Everolimus 5mg Daily | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
Number analyzed (Participants) | 6 | 7 | 11 | 35 | 19
score on a scale
  Baseline: number analyzed (Participants) | 4 | 5 | 9 | 34 | 19
  Baseline | 3.9 (1.4) | 1.3 (0.9) | 1.5 (1.2) | 2.0 (1.2) | 1.3 (0.9)
  Cycle 1: number analyzed (Participants) | 3 | 7 | 10 | 25 | 17
  Cycle 1 | 3.8 (1.0) | 1.6 (1.5) | 2.2 (1.8) | 2.5 (1.5) | 1.8 (1.2)
  Cycle 2: number analyzed (Participants) | 2 | 2 | 5 | 7 | 9
  Cycle 2 | 3.5 (1.3) | 1.9 (1.4) | 2.3 (1.7) | 3.4 (1.4) | 1.5 (1.3)
  Cycle 4: number analyzed (Participants) | 0 | 1 | 2 | 2 | 6
  Cycle 4 |  | 0.4 (0) | 1.3 (0.7) | 3.5 (2.1) | 1.8 (1.2)
  Cycle 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Cycle 6 |  |  |  |  | 1.4 (1.4)
  Cycle 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
  Cycle 8 |  |  |  |  | 1.8 (1.5)
  Cycle 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Cycle 10 |  |  |  |  | 1.5 (1.2)
  Cycle 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  Cycle 12 |  |  |  |  | 1.4 (1.0)

10. Secondary Outcome: Rate of Participants Symptom Interference With Function
Description: To evaluate the occurrence of symptoms and correlate to disease progression and tolerance to treatment using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) self-reporting tool. The MDASI-BT consists of 23 symptoms rated on an 11-point scale (0 - did not interfere, to 10 - interfered completely) to indicate the symptoms that interfere with a participant's life in the last 24 hours. We calculated the mean symptom interference at the time of clinical evaluation.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase I Dose Level I Sorafenib 400mg Twice Daily + Everolimus 5mg Daily | Phase I Dose Level -1 Sorafenib 400mg Twice Daily, 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on 7 Off + Everolimus 5mg Daily | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
Number analyzed (Participants) | 6 | 7 | 11 | 35 | 19
score on a scale
  Baseline: number analyzed (Participants) | 4 | 5 | 9 | 34 | 19
  Baseline | 5.0 (2.7) | 1.5 (1.6) | 2.3 (2.3) | 3.4 (2.7) | 2.1 (2.6)
  Cycle 1: number analyzed (Participants) | 3 | 7 | 10 | 25 | 17
  Cycle 1 | 4.2 (3.7) | 2.3 (2.4) | 3.3 (2.9) | 4.1 (2.8) | 2.5 (2.3)
  Cycle 2: number analyzed (Participants) | 2 | 2 | 5 | 7 | 9
  Cycle 2 | 5.0 (0.1) | 2.8 (3.7) | 4.3 (3.0) | 6.4 (2.2) | 1.8 (2.4)
  Cycle 4: number analyzed (Participants) | 0 | 1 | 2 | 2 | 6
  Cycle 4 |  | 0.3 (0) | 2.8 (3.1) | 4.2 (3.3) | 3.3 (3.2)
  Cycle 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Cycle 6 |  |  |  |  | 2.0 (2.8)
  Cycle 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3
  Cycle 8 |  |  |  |  | 2.4 (3.2)
  Cycle 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Cycle 10 |  |  |  |  | 1.6 (2.9)
  Cycle 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  Cycle 12 |  |  |  |  | 1.2 (1.6)

11. Other Pre Specified Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: A DLT is any grade 3 thrombocytopenia, grade 4 anemia, grade 4 neutropenia, or febrile neutropenia of any grade. Any non-hematologic grade 3 or grade 4 toxicity, excluding alopecia and/or hand/foot reaction. Failure to recover from toxicities (to grade 1 or less) to be eligible for re-treatment with sorafenib and everolimus within 14 days of the last dose of sorafenib and everolimus.
Time Frame: First 28 days of treatment only (cycle 1)
Population: Phase II is not applicable for this outcome measure. 6/7 subjects were evaluable in Dose Level-1 because one participant was excluded for under-dosing.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level I Sorafenib 400mg Twice Daily + Everolimus 5mg Daily | Phase I Dose Level -1 Sorafenib 400mg Twice Daily, 7 Days on, 7 Off + Everolimus 5mg Daily
Number analyzed (Participants) | 6 | 6
Participants | 3 | 1

12. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 21 months and 18 days, 30 months and twelve days, 83 months and 8 days, and 84 months and 26 days for each group respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level I Sorafenib 400mg Twice Daily + Everolimus 5mg Daily | Phase I Dose Level -1 Sorafenib 400mg Twice Daily, 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
Number analyzed (Participants) | 6 | 7 | 12 | 40 | 21
Participants | 6 | 7 | 12 | 38 | 20

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 21 months and 18 days, 30 months and twelve days, 83 months and 8 days, and 84 months and 26 days for each group respectively.
Arm/Group | Phase I Dose Level I Sorafenib 400mg Twice Daily + Everolimus 5mg Daily | Phase I Dose Level -1 Sorafenib 400mg Twice Daily, 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily
All-Cause Mortality (participants affected / at risk) | 5/6 | 6/7 | 9/12 | 19/40 | 11/21
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/7 | 3/12 | 12/40 | 2/21
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 12/12 | 38/40 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level I Sorafenib 400mg Twice Daily + Everolimus 5mg Daily (N=6) | Phase I Dose Level -1 Sorafenib 400mg Twice Daily, 7 Days on, 7 Off + Everolimus 5mg Daily (N=7) | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily (N=12) | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily (N=40) | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily (N=21)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Acute Sigmoid Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, altered mental status (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level I Sorafenib 400mg Twice Daily + Everolimus 5mg Daily (N=6) | Phase I Dose Level -1 Sorafenib 400mg Twice Daily, 7 Days on, 7 Off + Everolimus 5mg Daily (N=7) | Phase 2 Group A Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily (N=12) | Phase 2 Group B Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily (N=40) | Phase 2 Group C Dose Level -1 Sorafenib 400mg Twice Daily 7 Days on, 7 Off + Everolimus 5mg Daily (N=21)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0) | 2 (9) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2) | 5 (5) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood and lymphatic system disorders - Other, Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cholesterol high (Investigations) | 3 (4) | 3 (4) | 2 (2) | 7 (10) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (8) | 3 (4)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2) | 14 (18) | 6 (6)
Dizziness (Nervous system disorders) | 1 (3) | 1 (1) | 3 (3) | 3 (3) | 3 (3)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dysphasia (Nervous system disorders) | 2 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye disorders - Other, Left Homonymous Hemianopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, left peripheral vision loss (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, RIGHT HEMIANOPSIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, visual field deficit (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (5) | 4 (4) | 8 (12) | 15 (19) | 11 (15)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Gait disturbance (General disorders) | 3 (3) | 1 (2) | 1 (1) | 4 (4) | 1 (1)
Gastrointestinal disorders - Other, Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Epigastric Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Gas Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Loose Stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Loss of Appetite (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Insect Bite (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, Lip Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Onychocryptosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 5 (5) | 9 (11) | 7 (11)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (7) | 6 (7) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypersomnia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 1 (1) | 2 (4) | 12 (18) | 2 (5)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (5) | 3 (4) | 5 (5) | 6 (7) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 1 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Immune system disorders - Other, Right Underarm Abscess (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, MRSA pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Tinea Cruris (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Vaginal Yeast Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, Hypertriglyceridemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, Increased Total Bilirubin (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hyperlipidemia, may add statin to concomitant medications if continues to increase
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (6) | 1 (6) | 0 (0) | 8 (10) | 3 (8)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 2 (4)
Metabolism and nutrition disorders - Other, appetite decrease (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (4) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 5 (5) | 1 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Left Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4) | 9 (10) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Left wrist ganglio cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nervous system disorders - Other, Left Sixth Cranial Nerve Palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, Migraine headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, Pronator Drift Left Upper Extremity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, Unsteady Gait (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, cerebral edema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, right-sided numbness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (6)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Pain in extremity (General disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (3) | 3 (7) | 2 (4)
Papilledema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (4) | 1 (6) | 4 (5) | 9 (12) | 4 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Psychiatric disorders - Other, Dysphoric Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychiatric disorders - Other, Mood Alteration - Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 6 (11)
Respiratory, thoracic and mediastinal disorders - Other, Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 3 (8) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Left ear lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Rash, perianal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Rash; erythema annulare centrifugum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin and subcutaneous tissue disorders - Other, Right chest abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Skin sloughing (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, dry scalp (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, seborrheic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, under breasts, beginning on rt shoulder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, under breasts, groin area (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 2 (2)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 3 (3) | 1 (1) | 3 (3) | 4 (4) | 4 (9)

LIMITATIONS AND CAVEATS:
This study specifically addressed the question of whether the experimental regimen had benefit in the 2 important categories of recurrent glioblastoma: those who were bevacizumab treatment naive and those participants who had failed prior bevacizumab. Different efficacy metrics were used so that the "prior bevacizumab treatment arm" passed the Stage 1 of the 2-stage design, whereas the "bevacizumab naïve" did not. This is an important concept for future studies in recurrent glioblastoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT01434602/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT01434602/ICF_001.pdf